CLINICAL TRIAL: NCT02196285
Title: A Phase I, Open, Uncontrolled Study, to Evaluate the Safety and Imunogenicity of Double Viral Vaccine (MR) for Measles and Rubella in Young Adults
Brief Title: Study to Evaluate Safety and Imunogenicity of Double Viral Vaccine (MR) for Measles and Rubella
Acronym: MR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ASCLIN 002/2014
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Rubella; Measles
Keywords: Double; Viral; Vaccine; Measles; Rubella; Safety; Efficacy; Imunogenicity
MeSH Terms: conditions — Rubella; Measles | interventions — Vaccines; Rubella Vaccine; Measles Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Double viral vaccine (MR) (Experimental): Measles and rubella vaccine
  Interventions: Biological: Double viral (MR) vaccine

INTERVENTIONS:
Biological: Double viral (MR) vaccine — Measles and Rubella vaccine, as single arm
  Other Names: Measles and Rubella vaccine; MR Vaccine

SUMMARY:
Measles and rubella are highly contagious acute viral diseases. As per WHO, several evidences demonstrate the benefit for providing the universal access to vaccines containing measles and rubella antigens, mainly due to, respectively, mortality in children and malformations in fetuses. This is a Phase I, open study, non-controlled, to evaluate the safety, tolerability and imunogenicity of double viral vaccine anti-measles and rubella (MR), which is developed and produced at Instituto de Tecnologia em Imunobiologicos Bio-Manguinhos/Fiocruz, in Brazil, for use in human beings. 30 eligible volunteers, between 18-49 years old, will be vaccinated and monitored for local and systemic adverse events and titration of antibodies. The study will last 20 months in total.

DETAILED DESCRIPTION:
This is a Phase I, open study, non-controlled, to evaluate the safety, tolerability and imunogenicity of double viral vaccine anti-measles and rubella (MR), which is developed and produced at Instituto de Tecnologia em Imunobiologicos Bio-Manguinhos/Fiocruz, in Brazil, for use in human beings. 30 eligible volunteers, between 18-49 years old, will be vaccinated and monitored for local and systemic adverse events and titration of antibodies. The study will last 20 months in total.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 49 years old;
* Willing to provide name, address, telephone and other contact information in order to be contacted, whenever needed (example: in case of missing any scheduled visit, contact for confirmation of scheduling a visit, urgent safety notifications);
* Willing to strictly follow the study protocol;
* Capacity for understanding and signing in the Informed Consent Form;
* To understand the impossibility of participating in another clinical trial during the time of participation in the study, until 6 months after its conclusion;
* Intellectual level which allows to filling in the diaries for registering of symptoms at home;
* Willing to undergo to serological testing to HIV, HBV and HCV;
* Being in good health, with no significant medical history;
* Physical examination at screening period without clinically significant changes;
* Lab examination at screening period within the normal ranges, determined by the laboratory or abnormal values, grading below 1 or 2, according to medical decision.

Exclusion Criteria:

* Serious adverse reaction to any vaccination, as respiratory difficulty, angioedema and anaphylaxis;
* Acute or chronic disease, as diabetes, heart disease, systemic arterial hypertension;
* Use of anti-allergic with antigen injections in a maximum timeline of 14 days before the vaccination;
* Use of immunoglobulin in the past 12 months before the study vaccination;
* Use of blood products within 12 months before the vaccination;
* Use of any vaccine type within 30 days before the vaccination of the study;
* Chronic use of any medication, except homeopathy, and trivial ones, as nasal physiologic solution and vitamins;
* Previous immunosuppressive or cytotoxic medication, in the last 6 months. Individuals who have made use of this kind of medication in non-immunosuppressant doses, as nasal corticosteroid for allergic rhinitis of topic corticosteroid for non-complicated dermatitis, for more than 14 days, are allowed to be included in the study.
* Use of any kind of medication under investigation within one year before the vaccination.
* Unstable asthma or which may have required urgent care, hospitalization or intubation within the last 2 years, or which requires use of oral or intravenous corticosteroid.
* Coagulopathies diagnosed by a physician or report of capillary fragility (ex: bruises or bleedings without justifiable cause;
* Convulsions, except the ones caused by fever, before 2 years old;
* Psychiatric disease which difficults the adherence to the protocol, such as psychosis, obsessive-compulsive disorders, bipolar disease under treatment, diseases which require treatment with lithium and suicidal ideas in the last 5 years from the inclusion;
* Active malignant (p.e. any kind of cancer) or treated disease, to which the individual may relapse during the study;
* Asplenia (absence of spleen or its removal);
* Positive HIV in the screening examination of history of any immunosuppressant disease;
* Positive serology for C hepatitis in the screening evaluation;
* Positive Antigen HBs in the screening evaluation;
* Alcoholism (CAGE criteria), used for detection of abusive drinkers or alcoholic, validated in the Brazilian population with sensibility of 88% and specificity of 83%, if two or more answers, among four possible, are afirmative(Mansur and Monteiro, 1983), or according to medical decision;
* Abuse of illicit drugs, according to medical decision;
* Acquired or congenital immunodeficiency;
* Allergy to the vaccine compounds, as egg, neomycin and gelatin.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability analysis of the study vaccine | 9 months
  To evaluate the occurrence of serious adverse events among the subjects who have received study vaccine.

SECONDARY OUTCOMES:
Imunogenicity analysis | 9 months
  To evaluate imune response between post and pre-vaccination antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CerbinoNeto, PHD, Principal Investigator — Unidade de Ensaios Clínicos para Imunobiológicos, Fiocruz
Locations (1):
- Unidade de Ensaios Clínicos para Imunobiológicos, Rio de Janeiro, Rio de Janeiro, Brazil